CLINICAL TRIAL: NCT06826339
Title: A Multicenter, Prospective, Randomized Controlled Modified Multi-Platform (Matriarch) Trial Evaluating Several Cellular, Acellular, and Matrix-like Products (CAMPs) and Standard of Care Versus Standard of Care Alone in the Management of Nonhealing Diabetic Foot and Venous Leg Ulcers.
Brief Title: Evaluating Several Cellular, Acellular, and Matrix-like Products (CAMPs) and Standard of Care Versus Standard of Care Alone in the Management of Nonhealing Diabetic Foot and Venous Leg Ulcers.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tiger Biosciences, LLC. (Industry)
Collaborators: SerenaGroup, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TIGERCAMP
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Venous Leg Ulcer; Venous Leg; Diabetic Foot; Diabetic Foot Ulcer; Foot Ulcer, Diabetic; Ulcer Foot; Leg Ulcer; Ulcer Venous; Ulcer
MeSH Terms: conditions — Varicose Ulcer; Diabetic Foot; Foot Ulcer; Leg Ulcer; Ulcer | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: For a platform trial design, the allocation ratio is equal to the square root of the number of Intervention groups. This study will include 4 Intervention groups and 2 Control groups. A treatment effect of 0.35, significance level of 5%, 80% power, and a 1.4:1:1 for the VLU platform and 1.4:1:1 ratio for the DFU platform.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- DFU CAMP 1 + SOC = ACApatch™ + SOC (Experimental): ACApatch™ is a human amniotic membrane tissue allografts derived from human placental tissue.
  Interventions: Other: ACApatch™
- DFU CAMP 2 + SOC = caregraFT™ + SOC (Experimental): caregraFT™ is a human amniotic membrane tissue allografts derived from human placental tissue.
  Interventions: Other: caregraFT™
- DFU Standard of Care (Active Comparator): Standard of care will be cleaning, debridement, ulcer moisture balance, and offloading.
  Interventions: Other: Standard of Care
- VLU CAMP 1 + SOC = ACApatch™ + SOC (Experimental): ACApatch™ is a human amniotic membrane tissue allografts derived from human placental tissue.
  Interventions: Other: ACApatch™
- VLU CAMP 2 + SOC = caregraFT™ + SOC (Experimental): caregraFT™ is a human amniotic membrane tissue allografts derived from human placental tissue.
  Interventions: Other: caregraFT™
- VLU Standard of Care (Active Comparator): Standard of care will be cleaning, debridement, and ulcer moisture balance.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: ACApatch™ — Participants will receive weekly applications of ACApatch™ and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: DFU CAMP 1 + SOC = ACApatch™ + SOC; VLU CAMP 1 + SOC = ACApatch™ + SOC
Other: caregraFT™ — Participants will receive weekly applications of caregraFT™ and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: DFU CAMP 2 + SOC = caregraFT™ + SOC; VLU CAMP 2 + SOC = caregraFT™ + SOC
Other: Standard of Care — Beginning at the screening visit, participants will receive weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: DFU Standard of Care; VLU Standard of Care

SUMMARY:
Title A Multicenter, Prospective, Randomized Controlled Modified Multi-Platform (Matriarch) Trial Evaluating Several Cellular, Acellular, and Matrix-like Products (CAMPs) and Standard of Care versus Standard of Care alone in the Management of Nonhealing Diabetic Foot and Venous Leg Ulcers.

DETAILED DESCRIPTION:
To determine the between-arm difference in the proportion of subjects achieving complete closure of nonhealing diabetic foot ulcers and venous leg ulcers with multiple CAMPs plus SOC versus SOC alone over 12 weeks using a modified dual platform (Matriarch) trial design.

ELIGIBILITY:
Inclusion Criteria:(DFU)

* Subjects The potential subject must be at least 21 years of age or older.
* The potential subject must have a diagnosis of type 1 or 2 Diabetes mellitus.
* At enrollment, the potential subject must have a target ulcer with a minimum surface area of 1.0 cm2 and a maximum surface area of 20.0 cm2 measured post debridement.
* The potential subject must have a target ulcer that has been present for a minimum of 4 weeks and a maximum of 52 weeks of standard of care, prior to the initial screening visit.
* The potential subject must have a target ulcer located on the foot with at least 50% of the ulcer below the malleolus.
* The potential subject must have a target ulcer that is Wagner 1 or 2 grade, extending at least through the dermis or subcutaneous tissue and may involve the muscle provided it is below the medial aspect of the malleolus.
* The potential subject's affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 3 months of the first screening visit are acceptable:

  1. ABI between 0.7 and ≤ 1.3;
  2. TBI ≥ 0.6;
  3. TCOM ≥ 40 mmHg;
  4. PVR: biphasic.
* If the potential subject has two or more ulcers, they must be separated by at least 2 cm post-debridement. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer. The potential subject must have a target ulcers located on the plantar aspect of the foot must be offloaded for at least 14 days prior to enrollment.
* The potential subject must consent to using the prescribed offloading method for the duration of the study.
* The potential subject must agree to attend the weekly study visits required by the protocol.
* The potential subject must be willing and able to participate in the informed consent process.

Exclusion Criteria: (DFU)

* The potential subject is known to have a life expectancy of < 6 months.
* The potential subject's target ulcer is not secondary to diabetes.
* The potential subject's target ulcer is infected, requires systemic antibiotic therapy, or there is cellulitis in the surrounding skin.
* The potential subject's target ulcer exposes tendon or bone.
* There is evidence of osteomyelitis complicating the potential subject's target ulcer.
* The potential subject is receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of prednisone per day or equivalent) or cytotoxic chemotherapy or is taking medications that the PI believes will interfere with wound healing (e.g., biologics).
* The potential subject has applied topical steroids to the ulcer surface within one month of initial screening.
* The potential subject with a previous partial amputation on the affected foot that results in a deformity that impedes proper offloading of the target ulcer.
* The potential subject has glycated hemoglobin (HbA1c) greater than or equal to 12% within 3 months of the initial screening visit.
* The surface area of the potential subject's target ulcer has reduced in size by more than 20% in the 2 weeks prior to the initial screening visit ("historical" run-in period). EKare Imaging Device is not required for measurements taken during the historical run-in period (e.g., calculating surface area using length X width is acceptable).
* The surface area measurement of the potential subject's target ulcer decreases by 20% or more during the active 2-week screening phase: the 2 weeks from the initial screening visit (SV-1) to the TV-1 visit during which time the potential subject received SOC.
* The potential subject has an acute Charcot foot, or an inactive Charcot foot, which impedes proper offloading of the target ulcer.
* The potential subject is a woman who is pregnant or considering becoming pregnant within the next 6 months.
* The potential subject has end stage renal disease requiring dialysis.
* The potential subject has participated in a clinical trial involving treatment with an investigational product within the previous 30 days.
* A potential subject who, in the opinion of the investigator, has a medical or psychological condition that may interfere with study assessments.
* The potential subject was treated with hyperbaric oxygen therapy (HBOT) or a Cellular, Acellular, Matrix-like Product (CAMP) in the 30 days prior to the initial screening visit.
* The potential subject has a malnutrition indicator score <17 as measured on the Mini Nutritional Assessment.
* The potential subject has a wound with active or latent infection.
* The potential subject has a disorder that would create unacceptable risk of post-operative complication.

Inclusion Criteria:(VLU)

* The potential subject must be at least 21 years of age or older.
* At enrollment, the potential subjects must have a target ulcer with a minimum surface area of 1 cm2 and a maximum surface area of 20 cm2 measured post-debridement.
* The potential subject must have a target ulcer that has been present for a minimum of 4 weeks and a maximum of 52 weeks of standard of care prior to the initial screening visit.
* The potential subject has no visible signs of healing objectively, less than 40% reduction in wound size in the last 4 weeks.
* The potential subject's affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 3 months of the first screening visit are acceptable:

  1. ABI between 0.7 and ≤ 1.3;
  2. TBI ≥ 0.6;
  3. TCOM ≥ 40 mmHg;
  4. PVR: biphasic.
* If the potential subject has two or more ulcers, they must be separated by at least 2 cm post-debridement. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
* The potential subject must agree to attend the weekly study visits required by the protocol.
* The potential subject must be willing and able to participate in the informed consent process.

Exclusion Criteria: (VLU)

* The potential subject is known to have a life expectancy of < 6 months.
* The potential subject's target ulcer is infected, requires systemic antibiotic therapy, or there is cellulitis in the surrounding skin.
* The potential subject's target ulcer exposes tendon or bone.
* There is evidence of osteomyelitis complicating the potential subject's target ulcer.
* The potential subject is receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of prednisone per day or equivalent) or cytotoxic chemotherapy or is taking medications that the PI believes will interfere with wound healing (e.g., biologics).
* The potential subject has applied topical steroids to the ulcer surface within one month of initial screening.
* The potential subject has glycated hemoglobin (HbA1c) greater than or equal to 12% within 3 months of the initial screening visit.
* The surface area of the potential subject's target ulcer has reduced in size by more than 20% in the 2 weeks prior to the initial screening visit ("historical" run-in period). EKare Imaging Device is not required for measurements taken during the historical run-in period (e.g., calculating surface area using length X width is acceptable).
* The surface area measurement of the potential subject's target ulcer decreases by 20% or more during the active 2-week screening phase: the 2 weeks from the initial screening visit (SV-1) to the TV-1 visit during which time the potential subject received SOC.
* The potential subject is a woman who is pregnant or considering becoming pregnant within the next 6 months.
* The potential subject has end stage renal disease requiring dialysis.
* The potential subject has participated in a clinical trial involving treatment with an investigational product within the previous 30 days.
* A potential subject who, in the opinion of the investigator, has a medical or psychological condition that may interfere with study assessments.
* The potential subject was treated with hyperbaric oxygen therapy (HBOT) or a Cellular, Acellular, Matrix-like Product (CAMP) in the 30 days prior to the initial screening visit.
* The potential subject has a malnutrition indicator score <17 as measured on the Mini Nutritional Assessment.
* The potential subject has a wound with active or latent infection.
* The subject has a disorder that would create unacceptable risk of post-operative complication.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The between-arm difference in subjects that complete wound closure | 1-12 Weeks
  To determine the between-arm difference in the proportion of subjects achieving complete closure of nonhealing diabetic foot ulcers and venous leg ulcers with multiple CAMPs plus SOC versus SOC alone over 12 weeks using a modified dual platform (Matriarch) trial design. The platform design permits the inclusion of additional products by amending the protocol.

SECONDARY OUTCOMES:
Difference between CAMP plus SOC versus SOC alone in subjects that complete wound closure | 1-12 weeks
  To determine the between-arm difference in the time to closure over 12 weeks for CAMP plus SOC versus SOC alone.
Percent Area Reduction | 1-12 weeks
  To determine the between-arm difference in the percent area reduction (PAR) at weekly intervals the CAMP plus SOC arms versus SOC alone.
VAS | 1-12 Weeks
  To determine the between-arm difference in pain for patients that present with a VAS score of greater than 4.
Adverse Events | 1-12 weeks
  To evaluate the between-arm difference in the frequency and nature of adverse events in subjects receiving CAMP plus SOC versus SOC alone.

OTHER OUTCOMES:
Wound Quality of Life | 1-12 weeks
  To evaluate the between-arm difference in the quality of life for subjects receiving CAMP plus SOC compared to SOC alone using the Forgotten Wound Score (FWS) at treatment visits 1, 4, 8, and 12.
Wound Quality of Life | 1-12 weeks
  To evaluate the between-arm difference in the quality of life for subjects receiving CAMP plus SOC compared to SOC alone using the standard Wound Quality of Life (wQOL) questionnaires at treatment visits 1, 4, 8, and 12.
Age | 1-12 weeks
  To determine the proportion of ulcers that close in patients 65 years or older for CAMP plus SOC versus SOC alone.
Functional Ambulatory Category Scale | 1-12 weeks
  3. To evaluate the between-arm difference in functional ambulation based on Functional Ambulatory Category Scale (FACS) - VLU subjects only.

CONTACTS AND LOCATIONS:
Locations (1):
- Serena Group, Monroeville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No